CLINICAL TRIAL: NCT04726956
Title: A Combination of AKR1B10 and CA19-9 Improves the Diagnosis of Pancreatic Ductal Adenocarcinoma：A Multicenter Study
Brief Title: A Combination of AKR1B10 and CA19-9 Improves the Diagnosis of PDAC
Status: Completed | Type: Observational
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Lin Zhong, Director of Hepatobiliary and Pancreatic Surgery, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Other Study IDs: SHLTQC-3
Record Dates: First submitted 2021-01-26; First posted 2021-01-27 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2022-07

CONDITIONS: Pancreatic Ductal Adenocarcinoma
Keywords: pancreatic ductal adenocarcinoma; CA199; AKR1B10

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- case cohort: Pancreatic ductal adenocarcinoma patients (140)
- control cohort: healthy donors (140)
- Benign cohort: patients with Intraductal papillary mucinous tumor of the pancreas (IPMN), mucinous cystadenoma, or pancreatic cyst (30)

SUMMARY:
The purpose of this study is to clarify the diagnostic significance of AKR1B10 in patients with pancreatic ductal adenocarcinoma, and to combine with CA19-9 to improve the diagnosis rate of pancreatic ductal adenocarcinoma.

ELIGIBILITY:
General Inclusion Criteria

1. Age ≥ 18 years old;
2. Sign the informed consent form voluntarily;
3. Not a patient in the intensive care unit;

2. Patients with pancreatic ductal adenocarcinoma (PDAC group)

1. Two or more imaging studies (ultrasound, CT, MRI) found pancreatic tumors before operation, after surgical resection, intraoperative frozen pathology and postoperative pathology were clearly diagnosed as PDAC by 2 experienced pathologists, or diagnosed as pancreatic ductal adenocarcinoma by preoperative needle biopsy；
2. No other treatments such as radiotherapy or chemotherapy have been taken before the operation.

3. Benign disease group (Benign group)

1. Diagnosis of pancreatic intraductal papillary mucinous tumor (IPMN), mucinous cystadenoma or pancreas cyst based on clinical manifestations, clinical examinations, medical imagings (ultrasound/CT/MRI/ERCP), biopsy, and pathology
2. No relevant surgical treatment;

4. Healthy donors (Healthy group)

1. Healthy donors undergoing medical examinations at the above research centers;
2. Healthy donors of similar age without any benign or malignant diseases.

Exclusion Criteria:

1. PDAC group:

1. Patients who have undergone radiotherapy, chemotherapy and other tumor-related treatments before surgery;
2. Patients with non-primary pancreatic cancer;
3. Patients undergoing secondary operations;
4. Infected with HIV or AIDS related diseases;
5. Diagnosed as chronic or acute gastroenteritis;
6. Pregnant women;
7. Other situations that are not suitable for this research; 2. Benign group

(1) Patients who have undergone related surgical treatment in other hospitals; (2) Patients with a history of malignant tumors; 3. Healthy group:

1. Patients with a history of tumor;
2. Tumors found in medical examinations;
3. History of hepatitis B or C;
4. A history of acute or chronic gastroenteritis, cholecystitis, and cholangitis.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The population included in the case group was patients with clinically and pathologically clear pancreatic ductal adenocarcinoma; and the population included in the benign group was patients with clinically and pathologically clear IPMN, mucinous cystadenoma, or pancreas cyst; and the population included in the control group was a healthy population without any benign or malignant diseases.
Sampling Method: Non-Probability Sample
Enrollment: 258 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
CA199 and AKR1B10 were detected in the sera of PDAC patients and Benign patients before surgery, as well as in the sera of healthy donors | 1 week

SECONDARY OUTCOMES:
CA125, CEA, and AFP were detected in the sera of PDAC and Benign patients before surgery, as well as in the sera of healthy donors | 1 week

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Changhai Hospital of Shanghai, Shanghai
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou

IPD SHARING:
Plan to Share IPD: No